CLINICAL TRIAL: NCT04269304
Title: Deciphering AMD by Deep Phenotyping and Machine Learning- Prospective Study - PINNACLE
Acronym: PINNACLE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: Imperial College London (Other); University of Basel (Other); Medical University of Vienna (Other); University of Michigan (Other); King's College London (Other); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS - 256931; 47270 (Other: Sponsor Reference Number - University of Southampton); 210572/Z/18/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA for genotype analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Intermediate Age-Related Macular Degeneration Patients

SUMMARY:
We will conduct a prospective non-interventional study including 400 early AMD patients (=600 untreated early AMD eyes, including both unilateral (AREDS IV) and bilateral (≥AREDS II)) over a minimum of 1 year to specifically investigate the morphological sequence of events preceding the conversion towards late AMD. All patients will be followed by Optical Coherence Tomography (OCT) imaging every 4 months to detect the earliest focal sites of disease progression. As soon as focal areas of change are observed by the Vienna Reading Center (VRC), a targeted follow-up schedule will be triggered to investigate the events at that area of change in a targeted manner.

DETAILED DESCRIPTION:
We will recruit patients with 1) intermediate AMD in one eye and advanced AMD in the non-study eye or 2) patients with bilateral intermediate AMD (where both eyes will be included). As some participants are symptomless at the stage of intermediate AMD, we will recruit from hospital databases including imaging databases and ophthalmology and optometry practices and engagement with Patient Societies e.g. the Macular Society and patient public involvement meetings.

There will be four clinical sites performing detailed assessments on 50 patients each and, to increase sample size, an additional eight referral sites in the United Kingdom who will each enrol and follow 25 study patients by Spectral Domain Optical Coherence Tomography (SD-OCT) every 4 months. The acquired images from these referral sites will be sent to the Vienna Reading Centre for morphological identification of focal events. If a focal event is detected, participants will then be referred for a detailed, targeted assessment at either the University of Southampton or Moorfields Eye Hospital as detailed below.

After consent, patients will undergo visual function tests (ETDRS visual acuity, microperimetry) and multimodal imaging including fundus photographs, OCT scans, OCT angiography, autofluorescence and adaptive optics imaging. The visual function tests will be repeated annually and the multimodal imaging will be done at 4 monthly intervals for a minimum of 1 year. Blood will be taken within the first year for DNA analysis.

200 patients (main cohort) will undergo dense retinal phenotyping at a minimum of 4 visits.

Medical and smoking history, genotype and body mass index will also be included in the analysis as has been done previously. As well as structural tests, functional tests will be performed at baseline and end of the study using both microperimetry (a type of visual field test to create a "retinal sensitivity map" of the quantity of light perceived in specific parts of the retina) to identify focal changes and low luminance visual acuity to assess global changes. To increase sample size but make the study feasible an additional 200 patients at UK referral sites will undergo 4 monthly OCT and be referred to Southampton / Moorfields for dense phenotyping only if a focal event is detected by OCT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 55 years with either intermediate AMD (as defined by Ferris et al PMID: 23332590) in both eyes, i.e. large drusen > 125 um and/or any definite hyper- or hypopigmentary abnormalities associated with medium or large drusen; or intermediate AMD as defined above in one eye (study eye) and advanced AMD (geographic atrophy or choroidal neovascularization secondary to AMD) in the other eye.
* Subjects should have media clarity and pupillary dilation for adequate imaging and functional tests.

Exclusion Criteria:

* Co-existent ocular disease, which might affect visual function or retinal morphology
* Established glaucoma in either study eye or fellow eye with evidence of visual field loss or retinal nerve fibre loss (ocular hypertension is not an exclusion criterion unless associated with visual field loss or retinal nerve fibre loss in either eye).
* Cataract sufficient to affect retinal imaging
* Myopia > minus 6 diopters or a history of myopia > minus 6 diopters if patient has had cataract / refractive surgery.
* Major ocular surgery 3 months prior or anticipated within the next 6 months following enrolment.
* Taking drugs known to cause retinal toxicity such as hydroxychloroquine or tamoxifen
* OCT evidence of geographic atrophy (or complete Retinal Pigment Epithelium (RPE) and outer retinal atrophy (cRORA). This is (1) a region of hypertransmission of at least 250 mm in diameter, (2) a zone of attenuation or disruption of the RPE of at least 250 mm in diameter, (3) evidence of overlying photoreceptor degeneration, and (4) absence of scrolled RPE or other signs of an RPE tear.
* OCT evidence of choroidal neovascularization e.g sub-retinal scar tissue, sub-retinal fluid or intra-retinal fluid associated with a pigment epithelial detachment

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 1) intermediate AMD in one eye and advanced AMD in the non-study eye or 2) patients with bilateral intermediate AMD (where both eyes will be included).
Sampling Method: Non-Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity / specificity of OCT and autofluorescence parameters. | 3 years
  Identified by machine learning (ML) at predicting disease progression defined as focal conversion towards advanced AMD e.g. change in drusen volume, development of new geographic atrophy / choroidal neovascularisation.

SECONDARY OUTCOMES:
Sensitivity / specificity of novel imaging characteristics | 3 years
  For example, Adaptive Optics OCT (AO-OCT), OCT-A, at predicting disease progression; Receiver Operating Characteristic (ROC) curves; time from development of imaging change to development of these end-points; structure-function correlation; structure-genotype correlation; predictive risk models.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Lotery, Prof, Principal Investigator — University of Southampton
Locations (12):
- Medical University of Vienna, Vienna, Austria
- University Hospital Basel, Basel, Switzerland
- United Kingdom (10):
  - The Princess Alexandra Hospital Nhs Foundation Trust, Harlow, Essex
  - University Hospital Southampton, Southampton, Hampshire
  - St Mary's Hospital, Newport, Isle Of Wight
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Frimley Health Nhs Foundation Trust, Frimley, Surrey
  - Salisbury Nhs Foundation Trust, Salisbury, Wiltshire
  - University Hospitals Bristol and Weston Nhs Foundation Trust, Bristol
  - Moorfields Eye Hospital, London
  - Guy'S and St Thomas' Nhs Ft, London
  - St Mary's Hospital, Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Requests to access anonymised Individual Participant Data (IPD) can be made on application to the Trial Management Group Data Access Committee.
Supporting Information: Study Protocol, SAP
Time Frame: Currently available and can be accessed indefinitely.
Access Criteria: Requests for further information such as a clinical study report will be considered by the investigators following the end of the study and publication of primary outputs.
URL: https://pubmed.ncbi.nlm.nih.gov/35614343/

REFERENCES:
- [Derived] Anders P, Traber GL, Pfau M, Riedl S, Hagag AM, Camenzind H, Mai J, Kaye R, Bogunovic H, Fritsche LG, Rueckert D, Schmidt-Erfurth U, Sivaprasad S, Lotery AJ, Scholl HPN. Comparison of Novel Volumetric Microperimetry Metrics in Intermediate Age-Related Macular Degeneration: PINNACLE Study Report 3. Transl Vis Sci Technol. 2023 Aug 1;12(8):21. doi: 10.1167/tvst.12.8.21. PMID 37624605
- See also: Opt-out of PINNACLE (Retrospective) — https://clinicalresearch.uhs.nhs.uk/take-part
- See also: Protocol and statistical analysis plan PMID: 35614343 — https://pubmed.ncbi.nlm.nih.gov/35614343/